CLINICAL TRIAL: NCT03695354
Title: Impact of Whole-body Vibration Training on Sarcopenia in Geriatric Hospitalized Patients
Brief Title: Impact of Whole-body Vibration Training on Sarcopenic Elderly
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Jae-Young Lim, Professor, Department of Rehabilitation Medicine, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: B1607354003
Record Dates: First submitted 2018-10-02; First posted 2018-10-04 (Actual); Last update posted 2021-01-15 (Actual); Status verified 2021-01

CONDITIONS: Sarcopenia
Keywords: sarcopenia; vibration; gait; muscle; rehabilitation
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Whole body vibration plus conventional therapy group (Experimental): conventional therapy + whole body vibration training for 40 minutes per day, five days per week for two-week period.
  Interventions: Device: whole body vibration plus conventional therapy
- conventional training group (Active Comparator): conventional therapy (passive range of motion exercise and walking exercise) for 40 minutes per day, five days per week for two-week period.
  Interventions: Procedure: conventional therapy

INTERVENTIONS:
Device: whole body vibration plus conventional therapy — Subjects enrolled in whole body vibration training group are exposed to side-to-side alternating vertical sinusoidal vibration. Galileo system(Novotec Medical GmbH, Pforzheim, Germany) is used to training. Frequency of whole body vibration is 12Hz and amplitude is 4mm. After 10 minutes of vibration training, subjects rest 3 minutes. Then, additional 10 minutes of training will be given.
  conventional physical therapy is consisted of passive range of motion exercise and walking exercise.
  Arms: Whole body vibration plus conventional therapy group
Procedure: conventional therapy — conventional physical therapy is consisted of passive range of motion exercise and walking exercise.
  Arms: conventional training group

SUMMARY:
Sarcopenia is defined as a phenomenon which the amount of muscle mass in elderly aged 60-70 years is about 20-30% lower than that of the young adults and middle-aged people due to muscle atrophy caused by aging and alteration in muscle itself in aged skeletal muscle. Whole body vibration(WBV) training can be a choice for hospitalized patients who cannot conduct high intensity resistance training.

DETAILED DESCRIPTION:
This study is prospective study.

The goal of this study is

1. To investigate the effect of whole body vibration training using vibration platform with tilt table on muscle mass, muscle strength, physical performance in hospitalized older adults with sarcopenia.
2. To demonstrate whether whole body vibration training using vibration platform with tilt table can be useful in hospitalized older adults with sarcopenia who could not perform high intensity exercise.

ELIGIBILITY:
Inclusion Criteria:

* More than 70-year old people who admitted Seoul National University hospital, Bundang.
* Deconditioning subjects with diabetics, infections, chronic lung disease, etc. who cannot walk independently due to long-term hospital care.
* Subjects who had a mobility impairment.
* Subjects who can agree voluntarily.

Exclusion Criteria:

* Subjects who inserted implant due to trauma within 1~2 months recently.
* Acute coronary syndrome.
* Uncontrolled hypertension.
* Subjects who took drugs which can affects neuromuscular system.
* Severely impaired cognition
* Subjects who cannot agree volun.tarily.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-02-08 (Actual); Primary Completion 2021-05-31 (Estimated); Study Completion 2021-07-31 (Estimated)

PRIMARY OUTCOMES:
Berg balance scale | Before intervention / after two weeks intervention
  Change from baseline Berg balance scale to 2 weeks after initial assessment.
  Berg balance scale [from 0 to 56 score] is widely used to assess subjects' ability to control body balance.
  For '0' score, it means subject cannot maintain his/her own standing balance. For '56' score, he/she can properly keep static/dynamic standing balance.

SECONDARY OUTCOMES:
Maximal voluntary isometric contraction at knee | Before intervention / after two weeks intervention
  Change from baseline knee extension power to 2 weeks after initial assessment.
  Using the machine(muscle tester(manual), Lafayett instrument, USA), knee extension power will be measured while subject sit in the chair.
10 meter walking test | Before intervention / after two weeks intervention
  Change from baseline time when performing 10 meter walking test to 2 weeks after initial assessment.
  The subject was asked to move 10 meter away from baseline. While subject moved, total amount of time was measured. Then, the time used in first 2 meter movement and last time used in last 2 meter movement was excluded. Finally, total time used in 6 meter movement was measured.
Hand grip muscle strength | Before intervention / after two weeks intervention
  Change from baseline hand grip strength to 2 weeks after initial assessment.
  Its assessment is made by Leonardo Mechanograph(Novotec Medical GmbH, Pforzheim, Germany), (unit = N ). For the actual testing procedure, grip strength measurements of the bilateral limb were conducted. The subject was instructed to slowly squeeze the machine. Each measure site was tested one times during 3 seconds. The subjects sit in the chair, maintaining elbow flexed at 90 degree.

CONTACTS AND LOCATIONS:
Overall Officials: Jae-Young Lim, Ph.D., Study Director — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Verschueren SM, Bogaerts A, Delecluse C, Claessens AL, Haentjens P, Vanderschueren D, Boonen S. The effects of whole-body vibration training and vitamin D supplementation on muscle strength, muscle mass, and bone density in institutionalized elderly women: a 6-month randomized, controlled trial. J Bone Miner Res. 2011 Jan;26(1):42-9. doi: 10.1002/jbmr.181. PMID 20648661
- [Background] Santin-Medeiros F, Garatachea Vallejo N. [Musculoskeletal effects of vibration training in the elderly]. Rev Esp Geriatr Gerontol. 2010 Sep-Oct;45(5):281-4. doi: 10.1016/j.regg.2010.04.001. Epub 2010 May 23. Spanish. PMID 20546975
- [Background] von Stengel S, Kemmler W, Engelke K, Kalender WA. Effect of whole-body vibration on neuromuscular performance and body composition for females 65 years and older: a randomized-controlled trial. Scand J Med Sci Sports. 2012 Feb;22(1):119-27. doi: 10.1111/j.1600-0838.2010.01126.x. Epub 2010 May 24. PMID 20500555
- [Background] Kemmler W, V Stengel S, Mayer S, Niedermayer M, Hentschke C, Kalender WA. [Effect of whole body vibration on the neuromuscular performance of females 65 years and older. One-year results of the controlled randomized ELVIS study]. Z Gerontol Geriatr. 2010 Apr;43(2):125-32. doi: 10.1007/s00391-009-0074-0. Epub 2009 Oct 1. German. PMID 19789832
- [Background] Pietrangelo T, Mancinelli R, Toniolo L, Cancellara L, Paoli A, Puglielli C, Iodice P, Doria C, Bosco G, D'Amelio L, di Tano G, Fulle S, Saggini R, Fano G, Reggiani C. Effects of local vibrations on skeletal muscle trophism in elderly people: mechanical, cellular, and molecular events. Int J Mol Med. 2009 Oct;24(4):503-12. doi: 10.3892/ijmm_00000259. PMID 19724891
- [Background] Machado A, Garcia-Lopez D, Gonzalez-Gallego J, Garatachea N. Whole-body vibration training increases muscle strength and mass in older women: a randomized-controlled trial. Scand J Med Sci Sports. 2010 Apr;20(2):200-7. doi: 10.1111/j.1600-0838.2009.00919.x. Epub 2009 Apr 20. PMID 19422657
- [Background] Kaeding TS. [Sarcopenia and whole body vibration training: an overview]. Z Gerontol Geriatr. 2009 Apr;42(2):88-92. doi: 10.1007/s00391-008-0565-4. Epub 2008 Aug 29. German. PMID 18726053
- [Background] Bogaerts A, Delecluse C, Claessens AL, Coudyzer W, Boonen S, Verschueren SM. Impact of whole-body vibration training versus fitness training on muscle strength and muscle mass in older men: a 1-year randomized controlled trial. J Gerontol A Biol Sci Med Sci. 2007 Jun;62(6):630-5. doi: 10.1093/gerona/62.6.630. PMID 17595419
- [Background] Cardinale M, Rittweger J. Vibration exercise makes your muscles and bones stronger: fact or fiction? J Br Menopause Soc. 2006 Mar;12(1):12-8. doi: 10.1258/136218006775997261. PMID 16513017
- [Background] Cardinale M, Wakeling J. Whole body vibration exercise: are vibrations good for you? Br J Sports Med. 2005 Sep;39(9):585-9; discussion 589. doi: 10.1136/bjsm.2005.016857. PMID 16118292
- [Background] Cardinale M, Pope MH. The effects of whole body vibration on humans: dangerous or advantageous? Acta Physiol Hung. 2003;90(3):195-206. doi: 10.1556/APhysiol.90.2003.3.2. PMID 14594190
- [Background] Roelants M, Delecluse C, Verschueren SM. Whole-body-vibration training increases knee-extension strength and speed of movement in older women. J Am Geriatr Soc. 2004 Jun;52(6):901-8. doi: 10.1111/j.1532-5415.2004.52256.x. PMID 15161453
- [Background] Rees S, Murphy A, Watsford M. Effects of vibration exercise on muscle performance and mobility in an older population. J Aging Phys Act. 2007 Oct;15(4):367-81. doi: 10.1123/japa.15.4.367. PMID 18048942
- [Background] Rees SS, Murphy AJ, Watsford ML. Effects of whole body vibration on postural steadiness in an older population. J Sci Med Sport. 2009 Jul;12(4):440-4. doi: 10.1016/j.jsams.2008.02.002. Epub 2008 Jun 11. PMID 18550436
- [Background] Jordan MJ, Norris SR, Smith DJ, Herzog W. Vibration training: an overview of the area, training consequences, and future considerations. J Strength Cond Res. 2005 May;19(2):459-66. doi: 10.1519/13293.1. PMID 15903391
- [Background] Cheung WH, Mok HW, Qin L, Sze PC, Lee KM, Leung KS. High-frequency whole-body vibration improves balancing ability in elderly women. Arch Phys Med Rehabil. 2007 Jul;88(7):852-7. doi: 10.1016/j.apmr.2007.03.028. PMID 17601464
- [Background] Song GE, Kim K, Lee DJ, Joo NS. Whole body vibration effects on body composition in the postmenopausal korean obese women: pilot study. Korean J Fam Med. 2011 Nov;32(7):399-405. doi: 10.4082/kjfm.2011.32.7.399. Epub 2011 Nov 30. PMID 22745878
- [Background] Park YG, Kwon BS, Park JW, Cha DY, Nam KY, Sim KB, Chang J, Lee HJ. Therapeutic effect of whole body vibration on chronic knee osteoarthritis. Ann Rehabil Med. 2013 Aug;37(4):505-15. doi: 10.5535/arm.2013.37.4.505. Epub 2013 Aug 26. PMID 24020031
- [Background] Lee BK, Chon SC. Effect of whole body vibration training on mobility in children with cerebral palsy: a randomized controlled experimenter-blinded study. Clin Rehabil. 2013 Jul;27(7):599-607. doi: 10.1177/0269215512470673. Epub 2013 Feb 14. PMID 23411791
- [Background] Smoliner C, Sieber CC, Wirth R. Prevalence of sarcopenia in geriatric hospitalized patients. J Am Med Dir Assoc. 2014 Apr;15(4):267-72. doi: 10.1016/j.jamda.2013.11.027. PMID 24679831
- [Background] Patel HP, Syddall HE, Jameson K, Robinson S, Denison H, Roberts HC, Edwards M, Dennison E, Cooper C, Aihie Sayer A. Prevalence of sarcopenia in community-dwelling older people in the UK using the European Working Group on Sarcopenia in Older People (EWGSOP) definition: findings from the Hertfordshire Cohort Study (HCS). Age Ageing. 2013 May;42(3):378-84. doi: 10.1093/ageing/afs197. Epub 2013 Feb 5. PMID 23384705
- [Background] Kim IH. Age and gender differences in the relation of chronic diseases to activity of daily living (ADL) disability for elderly South Koreans: based on representative data. J Prev Med Public Health. 2011 Jan;44(1):32-40. doi: 10.3961/jpmph.2011.44.1.32. PMID 21483221